CLINICAL TRIAL: NCT02739815
Title: Comparative Study For Role Of Different Prophylactic Doses Of Intravenous Tranexamic Acid In Reducing Blood Loss At Caesarean Section: A Randomised Controlled Trial
Brief Title: Role Of Different Prophylactic Doses Of Intravenous Tranexamic Acid In Reducing Blood Loss At Caesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Talkha Central Hospital (Other Government)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Amro Mohamed Ibrahim Ibrahim Hetta, Master Degree Student of Obstetrics and Gynecology, Al-Azhar University, Talkha Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OG1
Record Dates: First submitted 2016-04-04; First posted 2016-04-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Hemorrhage of Cesarean Section and/or Perineal Wound; Postpartum Hemorrhage
Keywords: Caesarean Section; Tranexamic Acid; Postpartum Hemorrhage; Ecbolics
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Will receive a placebo (10 ml of distilled water) in Z solution [500 ml of normal saline containing a prophylactic Antibiotic 1 g] (At 20 minutes preoperatively).
  Interventions: Drug: Normal Saline containing a prophylactic Antibiotic 1 g
- T1 (Active Comparator): Will receive Tranexamic acid 15 mg/kg in Z solution [500 ml of normal saline containing a prophylactic Antibiotic 1 g] (At 20 minutes preoperatively).
  Interventions: Drug: Normal Saline containing a prophylactic Antibiotic 1 g; Drug: Tranexamic Acid
- T2 (Active Comparator): Will receive Tranexamic acid 20 mg/kg in Z solution [500 ml of normal saline containing a prophylactic Antibiotic 1 g] (At 20 minutes preoperatively).
  Interventions: Drug: Normal Saline containing a prophylactic Antibiotic 1 g; Drug: Tranexamic Acid
- T3 (Active Comparator): Will receive Tranexamic acid 25 mg/kg in Z solution [500 ml of normal saline containing a prophylactic Antibiotic 1 g] (At 20 minutes preoperatively).
  Interventions: Drug: Normal Saline containing a prophylactic Antibiotic 1 g; Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Normal Saline containing a prophylactic Antibiotic 1 g — 500 ml of normal saline containing a prophylactic Antibiotic 1 g.
  Other Names: Solution of Sodium Chloride 0.9 %
Drug: Tranexamic Acid — Tranexamic acid
  Other Names: TXA
  Arms: T1; T2; T3

SUMMARY:
This study aims to define a safe prophylactic intravenous TXA dose with an advantage over others in reducing total blood loss volume at secondary uncomplicated LSCS.

DETAILED DESCRIPTION:
Bleeding during vaginal or operative delivery is always of prime concern. Despite significant progress in obstetric care 125,000 women die from obstetric hemorrhage annually in the world.

The incidence of CS is increasing, and the average blood loss during CS (1000 mL) is double the amount lost during vaginal delivery (500 mL). CS rate as high as 25-30% in many areas of the world. In Egypt the CS rate is 27.6 %, in United States of America, from 1970-2009 the CS rate rose from 4.5-32.9%, and declined to 32.8% of all deliveries at 2010. In spite of the various measures to prevent blood loss during and after CS, post-partum hemorrhage (PPH) continues to be the most common complication seen in almost 20% of the cases, and causes approximately 25% of maternal deaths worldwide, leading to increased maternal morbidity and mortality. Women who undergo a CS are much more likely to be delivered by a repeat operation in subsequent pregnancies. For women undergoing subsequent CS, the maternal risks are even greater like massive obstetric hemorrhage, hysterectomy, admission to an intensive care unit, or maternal death. Medications, such as oxytocin, misoprostol and prostaglandin F2α, have been used to control bleeding postoperatively.

TXA is a synthetic analog of the amino acid lysine,10 as an antifibrinolytic agent it has roughly eight times the antifibrinolytic activity of an older analogue; ε-aminocaproic acid. It competitively inhibits the activation of plasminogen to plasmin, by binding to specific sites of both plasminogen and plasmin, a molecule responsible for the degradation of fibrin, a protein that forms the framework of blood clots. Its intravenous administration has been routinely used for many years to reduce or prevent excessive hemorrhage in various medical conditions or disorders (helping hemostasis), also during and after surgical procedures like benign hysterectomy, open heart surgeries, scoliosis surgery, oral surgery, liver surgeries, total hip or knee arthroplasty, and urology. It has been shown to be very useful and efficient in reducing blood loss and incidence of blood transfusion in these surgeries, and decreases the risk of death in bleeding trauma patients. It was also included in the World Health Organization (WHO) Model List of Essential Medicines.

About its role in CS, some recent studies showed that TXA has advantage and useful effect safely in reducing blood loss and requirement of additional ecbolics. Its doses used intravenously to reduce blood loss at CS were a bolus of 1gm, 10 mg/kg, or 15 mg/kg which had an advantage over 10 mg/kg in anemic parturients. No defined safe prophylactic intravenous TXA dose being found in searching literature having an advantage over other doses in reducing total blood loss especially at secondary uncomplicated LSCS.

ELIGIBILITY:
Inclusion Criteria:

* Maternal average age of 20-40 years.
* Singleton pregnancy at term between 38±5 days and 40 weeks.
* Elective planned or emergency secondary lower segment caesarean sections (LSCS).

Exclusion Criteria:

* Women with severe medical and surgical complications as any of the following will be excluded :

  * Heart, liver, kidney, or brain diseases, and blood disorders.
  * Abruptio placenta, and placental abnormalities or accrete syndromes.
  * Polyhydramnios, macrosomia, preeclampsia, or allergy to tranexamic acid.
  * History of thromboembolic disorders, or severe anemia.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Total Blood Loss Volume | Up to 7 hours
  Estimating Total Blood Loss Volume (ml) during and after Caesarean Section, up to 6 hours post-operative.

SECONDARY OUTCOMES:
Duration of surgery | Up to One hour
  Duration of Caesarean Section estimating (min)
Hemoglobin level (Hb) | 6 hours
  6 hours post-operative hemoglobin level (mg/dL) estimating.
Maternal weight (W) | 2 hours
  2 hours post-operative maternal weight (kg) estimating
Hematocrit value (Hct) | 6 hours
  6 hours post-operative hematocrit value (%) estimating.
Need for blood or blood products transfusion | Up to 6 hours
  Need for other medical measures to arrest and manage bleeding (transfusion of blood or blood products)
Need for additional ecbolics | Up to 6 hours
  Need for other medical measures to arrest and manage bleeding if there is a uterine atony (more than five units of intravenous Syntocinon®)
Need for hysterectomy | Up to 6 hours
  Need for other surgical measures to arrest and manage bleeding (Hysterectomy)
Need for uterine artery ligation | Up to 6 hours
  Need for other surgical measures to arrest and manage bleeding (Uterine artery ligation)
Need for B-lynch | Up to 6 hours
  Need for other surgical measures to arrest and manage bleeding if there is a uterine atony (B-lynch)
APGAR Score | Up to 30 minutes
  APGAR Score as index for any neonatal side effects of medications given
Any sign for developing a thromboembolic disorder (Maternal) | One week
  As index for any maternal side effects of medications given
Blood pressure | Up to 2 hours
  Measuring maternal blood pressure (mmHg) immediately postoperative and after 2 hours postoperative.
Pulse rate | Up to 2 hours
  Measuring maternal blood puse rate (/minute) immediately postoperative and after 2 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Amro M. Hetta, MS Student, Principal Investigator — Al-Azhar University, Faculty of Medicine for boys (Cairo), Departments of OBS/GYN; Mahmoud E. Mohammed, Professor, Study Director — Al-Azhar University, Faculty of Medicine for boys (Cairo), Departments of OBS/GYN; Yehia A. Wafa, Chairman, Study Chair — Al-Azhar University, Faculty of Medicine for boys (Cairo), Departments of OBS/GYN
Locations (1):
- Al-Azhar University, Faculty of Medicine for Boys ( Cairo ), Al-Hussein University Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martin JA, Hamilton BE, Ventura SJ, Osterman MJ, Wilson EC, Mathews TJ. Births: final data for 2010. Natl Vital Stat Rep. 2012 Aug 28;61(1):1-72. PMID 24974589
- [Background] Gungorduk K, Yildirim G, Asicioglu O, Gungorduk OC, Sudolmus S, Ark C. Efficacy of intravenous tranexamic acid in reducing blood loss after elective cesarean section: a prospective, randomized, double-blind, placebo-controlled study. Am J Perinatol. 2011 Mar;28(3):233-40. doi: 10.1055/s-0030-1268238. Epub 2010 Oct 26. PMID 20979013
- [Background] Cahill AG, Stamilio DM, Odibo AO, Peipert JF, Ratcliffe SJ, Stevens EJ, Sammel MD, Macones GA. Is vaginal birth after cesarean (VBAC) or elective repeat cesarean safer in women with a prior vaginal delivery? Am J Obstet Gynecol. 2006 Oct;195(4):1143-7. doi: 10.1016/j.ajog.2006.06.045. Epub 2006 Jul 17. PMID 16846571
- [Background] Marshall NE, Fu R, Guise JM. Impact of multiple cesarean deliveries on maternal morbidity: a systematic review. Am J Obstet Gynecol. 2011 Sep;205(3):262.e1-8. doi: 10.1016/j.ajog.2011.06.035. Epub 2011 Jun 15. PMID 22071057
- [Background] Silver RM, Landon MB, Rouse DJ, Leveno KJ, Spong CY, Thom EA, Moawad AH, Caritis SN, Harper M, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, Peaceman AM, O'Sullivan MJ, Sibai B, Langer O, Thorp JM, Ramin SM, Mercer BM; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Maternal morbidity associated with multiple repeat cesarean deliveries. Obstet Gynecol. 2006 Jun;107(6):1226-32. doi: 10.1097/01.AOG.0000219750.79480.84. PMID 16738145
- [Background] Yehia AH, Koleib MH, Abdelazim IA, Atik A. Tranexamic acid reduces blood loss during and after cesarean section: A double blinded, randomized, controlled trial. Asian Pacific Journal of Reproduction. 2014 Mar 31;3(1):53-6.
- [Background] Tarabrin O, Kaminskiy V, Galich S, Tkachenko R, Gulyaev A, Shcherbakov S, Gavrychenko D. Efficacy of tranexamic acid in decreasing blood loss during cesarean section. Critical Care. 2012;16(Suppl 1):P439.
- [Background] Mayur G, Purvi P, Ashoo G, Pankaj D. Efficacy of tranexamic acid in decreasing blood loss during and after cesarean section: a randomized case controlled prospective study. J Obstet Gynecol India. 2007;57(3):227-30.
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Movafegh A, Eslamian L, Dorabadi A. Effect of intravenous tranexamic acid administration on blood loss during and after cesarean delivery. Int J Gynaecol Obstet. 2011 Dec;115(3):224-6. doi: 10.1016/j.ijgo.2011.07.015. Epub 2011 Aug 27. PMID 21872857
- [Background] Ahmed MR, Sayed Ahmed WA, Madny EH, Arafa AM, Said MM. Efficacy of tranexamic acid in decreasing blood loss in elective caesarean delivery. J Matern Fetal Neonatal Med. 2015 Jun;28(9):1014-8. doi: 10.3109/14767058.2014.941283. Epub 2014 Jul 28. PMID 25068947
- [Background] Maged AM, Helal OM, Elsherbini MM, Eid MM, Elkomy RO, Dahab S, Elsissy MH. A randomized placebo-controlled trial of preoperative tranexamic acid among women undergoing elective cesarean delivery. Int J Gynaecol Obstet. 2015 Dec;131(3):265-8. doi: 10.1016/j.ijgo.2015.05.027. Epub 2015 Aug 15. PMID 26341174
- [Background] Wang HY, Hong SK, Duan Y, Yin HM. Tranexamic acid and blood loss during and after cesarean section: a meta-analysis. J Perinatol. 2015 Oct;35(10):818-25. doi: 10.1038/jp.2015.93. Epub 2015 Jul 30. PMID 26226243
- [Background] Goswami U, Sarangi S, Gupta S, Babbar S. Comparative evaluation of two doses of tranexamic acid used prophylactically in anemic parturients for lower segment cesarean section: A double-blind randomized case control prospective trial. Saudi J Anaesth. 2013 Oct;7(4):427-31. doi: 10.4103/1658-354X.121077. PMID 24348295
- [Background] Gibbons L, Belizán JM, Lauer JA, Betrán AP, Merialdi M, Althabe F. The global numbers and costs of additionally needed and unnecessary caesarean sections performed per year: overuse as a barrier to universal coverage. World health report 2010, 30: 1-31.
- [Background] WHO Recommendations for the Prevention and Treatment of Postpartum Haemorrhage. Geneva: World Health Organization; 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK131942/ PMID 23586122
- [Background] Shahid A, Khan A. Tranexamic acid in decreasing blood loss during and after caesarean section. J Coll Physicians Surg Pak. 2013 Jul;23(7):459-62. PMID 23823946
- [Background] Sentilhes L, Lasocki S, Ducloy-Bouthors AS, Deruelle P, Dreyfus M, Perrotin F, Goffinet F, Deneux-Tharaux C. Tranexamic acid for the prevention and treatment of postpartum haemorrhage. Br J Anaesth. 2015 Apr;114(4):576-87. doi: 10.1093/bja/aeu448. Epub 2015 Jan 8. PMID 25571934
- [Background] Gaines-Dillard N, Bartley MK, Rosini JM. Tranexamic acid in the trauma patient. Nursing. 2016 Feb;46(2):60-2. doi: 10.1097/01.NURSE.0000476234.78599.e2. No abstract available. PMID 26760392
- [Background] Topsoee MF, Bergholt T, Ravn P, Schouenborg L, Moeller C, Ottesen B, Settnes A. Anti-hemorrhagic effect of prophylactic tranexamic acid in benign hysterectomy-a double-blinded randomized placebo-controlled trial. Am J Obstet Gynecol. 2016 Jul;215(1):72.e1-8. doi: 10.1016/j.ajog.2016.01.184. Epub 2016 Jan 30. PMID 26829509
- [Background] Sujata N, Tobin R, Kaur R, Aneja A, Khanna M, Hanjoora VM. Randomized controlled trial of tranexamic acid among parturients at increased risk for postpartum hemorrhage undergoing cesarean delivery. Int J Gynaecol Obstet. 2016 Jun;133(3):312-5. doi: 10.1016/j.ijgo.2015.09.032. Epub 2016 Feb 16. PMID 26952346
- [Background] Simonazzi G, Bisulli M, Saccone G, Moro E, Marshall A, Berghella V. Tranexamic acid for preventing postpartum blood loss after cesarean delivery: a systematic review and meta-analysis of randomized controlled trials. Acta Obstet Gynecol Scand. 2016 Jan;95(1):28-37. doi: 10.1111/aogs.12798. Epub 2015 Nov 12. PMID 26698831
- [Background] Gupta A, Dwivedi Y, Shakya V, Srivastva U, Saxena A, Agarwal AM, et al. Efficacy of Tranexamic Acid in Reducing Perioperative Blood Loss During Caesarean Section: A Placebo Controlled Double Blind Study. International Journal of Scientific Research 2016, 5(3).
- [Background] Gai MY, Wu LF, Su QF, Tatsumoto K. Clinical observation of blood loss reduced by tranexamic acid during and after caesarian section: a multi-center, randomized trial. Eur J Obstet Gynecol Reprod Biol. 2004 Feb 10;112(2):154-7. doi: 10.1016/s0301-2115(03)00287-2. PMID 14746950
- [Background] Sekhavat L, Tabatabaii A, Dalili M, Farajkhoda T, Tafti AD. Efficacy of tranexamic acid in reducing blood loss after cesarean section. J Matern Fetal Neonatal Med. 2009 Jan;22(1):72-5. doi: 10.1080/14767050802353580. PMID 19165682